CLINICAL TRIAL: NCT00779402
Title: Autologous PAP-loaded Dendritic Cell Vaccine (Sipuleucel-T, APC8015, Provenge®) in Patients With Non-metastatic Prostate Cancer Who Experience PSA Elevation Following Radical Prostatectomy: a Randomized, Controlled, Double-blind Trial
Brief Title: PROvenge Treatment and Early Cancer Treatment
Acronym: PROTECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-11
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: cancer; prostate cancer; prostatectomy; PSA; sipuleucel-T; PROVENGE; APC8015; non-metastatic; nonmetastatic; androgen-sensitive; androgen sensitive; biochemical recurrence; biochemically recurrent; immune therapy; immunotherapy; vaccine; dendritic cells; antigen-presenting cells; antigen presenting cells; cancer vaccine; therapeutic vaccine; therapeutic cancer vaccine; biologic; booster
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sipuleucel-T (Experimental): Subjects received infusion of Sipuleucel-T, at 2-week intervals, for a total of 3 infusions.
  Interventions: Biological: Sipuleucel-T
- Control (Placebo Comparator): Subjects received infusion of control (autologous cellular product consisting of antigen presenting cells (APCs) prepared in the absence of PA2024 antigen) at 2-week intervals, for a total of 3 infusions.
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — Autologous cellular product consisting of antigen presenting cells (APCs) prepared in the absence of PA2024 antigen.
  Arms: Control
Biological: Sipuleucel-T — Sipuleucel-T is an autologous cellular product consisting of antigen presenting cells (APCs) activated with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  Other Names: Provenge®; APC8015
  Arms: Sipuleucel-T

SUMMARY:
The PROTECT-PROvenge Treatment and Early Cancer Treatment trial was a Phase III trial for patients with hormone sensitive prostate cancer. The study was conducted at over 15 participating centers throughout the US. The purpose of the study was to determine if sipuleucel-T was effective for treatment of early stage, non-metastatic prostate cancer. The study compared the active vaccine to control to determine whether the product delayed the time until cancer progression.

DETAILED DESCRIPTION:
This was a prospective, double blind, controlled, randomized trial of immunotherapy with prostatic acid phosphatase (PAP)-loaded autologous antigen presenting cells (APCs), in subjects with non metastatic prostate cancer. Subjects that qualified for this study were men who had previously undergone a prostatectomy and whose only sign of disease recurrence was a rise in serum prostate specific antigen (PSA).

The primary objectives were to compare the time to biochemical failure (BF, PSA greater than or equal to 3 ng/mL) between sipuleucel-T (treatment group) and control, and to study the safety of sipuleucel-T.

Following short-term open-label treatment with a luteinizing hormone-releasing hormone-analogue (LHRH-a), Subjects completed a checklist designed to compare androgen suppression-related side effects during periods with and without androgen suppression.

Subjects who achieved a PSA of < 1 ng/ml were randomized to blinded treatment assignments of either sipuleucel-T or control in a 2:1 ratio. Following randomization, subjects underwent 3 leukapheresis procedures on alternate weeks (Weeks 0, 2, and 4). Approximately three days following each leukapheresis procedure, subjects received an infusion of either sipuleucel-T or control.

At the time BF was confirmed, subjects were eligible for a booster infusion. The booster process consisted of 1 leukapheresis procedure followed by 1 infusion of sipuleucel-T. The booster process, in effect under protocol amendment 5, differed from the previous booster process that consisted of 1 infusion of the same treatment assigned at randomization (sipuleucel-T or control).

Subjects continued to be observed until DF was confirmed by bone scan or computed tomography (CT) scan, or other imaging modalities as clinically indicated. After confirmed DF, subjects were followed by telephone every 6 months for safety and survival, treatment-related AEs, any CVEs, or new therapies for prostate cancer.

ELIGIBILITY:
Inclusion Criteria for the Run-In Phase (Week -13)

* Histologic diagnosis of adenocarcinoma of the prostate.
* Within at least 3 months, but not more than 10 years, prior to initiation of the run-in phase with LHRH-a depot, the subject has undergone a radical prostatectomy for Stage T1b - T3c, N0 - N1, Nx, or M0 disease Subjects who experienced their first PSA recurrence within 2 years post completion of initial therapy of curative intent was eligible without consideration of the Gleason score of the tumor specimen. Subjects who experienced their first PSA relapse between 2 and 10 years post completion of initial therapy of curative intent was eligible only if the Gleason score of the tumor specimen was ≥ 7.
* Therapeutic PSA response to primary therapy was below 0.4 ng/mL.
* Tumor specimen positive for PAP.
* PSA relapse while not currently receiving androgen ablation therapy.
* If androgen ablation was given for a previous PSA relapse, PSA must have increased to a level at least 25% above the nadir observed while on this therapy, and to an absolute level of at least 3 ng/mL.
* Subjects who had been treated with adjuvant or salvage radiation following radical prostatectomy, or with either LHRH-a (e.g., leuprolide acetate or goserelin acetate) or non-steroidal anti-androgen therapy (e.g., bicalutamide 150 mg/day) for a prior PSA relapse, may enter the study provided: Post-prostatectomy PSA was never ≥ 20 ng/mL; PSA was not rising while subject received hormonal therapy, and; For any hormonal therapy received, the last effective day of androgen deprivation was at least 6 months prior to the date of LHRH-a depot placement.
* Confirmed Stage M0 disease.
* Estimated life expectancy of at least 1 year.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Ability to understand the trial procedures and requirements.
* ≥ 18 and ≤ 80 years of age.
* Ability to understand and willingness to sign an informed consent form.

Exclusion Criteria:

Exclusion Criteria for Entry into the Run-In Phase (Week -13)

* Metastasis.
* Clinical evidence of local recurrence other than PSA elevation (e.g., palpable induration or mass in the prostatic fossa).
* Any surgery within 4 weeks prior to the date of LHRH-a depot placement.
* Prior orchiectomy.
* PSA ≥ 20 ng/mL at any time after radical prostatectomy.
* Current systemic steroid therapy (inhaled or topical steroids are acceptable).
* Any chemotherapy within 4 months prior to the LHRH-a depot placement.
* Prior immunotherapy or therapy with other experimental agents for prostate cancer.
* Treatment with radioactive seeds within 12 months prior to the LHRH a depot placement.
* History of any other prior malignancy other than resected basal or squamous cell carcinoma of the skin within 5 years of entry.
* Concurrent participation in another clinical trial involving experimental medication.
* Any disease, condition, social, or geographical constraint that in the opinion of the Investigator or medical monitor reduced the probability that the subject will complete the trial or affects the evaluation of study end points

Exclusion Criteria for Randomization (Week 0):

* Central laboratory value of PSA ≥ 1 ng/mL at the end of the LHRH-a run-in phase.
* Randomized more than 3 weeks following the last effective date of testicular androgen suppression (as described in the package insert).
* Any use of herbal preparations (e.g., Prostate Cancer (PC) -SPES or saw palmetto) within 4 weeks prior to randomization.
* Any contraindication to leukapheresis or infusion of sipuleucel-T or control.
* Positive serology for human immunodeficiency virus (HIV)-1 or 2, human lymphotropic virus (HTLV)-1 or 2, or evidence of active Hepatitis B or C infection.
* Any ongoing active bacterial, viral, or fungal infection.

Exclusion Criteria During the Trial:

* The use of any systemic therapy for prostate cancer following randomization and prior to BF (PSA ≥ 3 ng/mL).
* Placement of radioactive seeds or salvage radiation before BF (PSA ≥ 3 ng/mL) documented.
* Initiation of systemic corticosteroids at doses greater than the equivalent of 40 mg hydrocortisone per day (inhaled steroids are allowed) before BF.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2001-10; Primary Completion 2006-08 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Israel, MD, Study Director — Valeant Pharmaceuticals North America LLC
Locations (18):
- United States (18):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - South Orange County Medical Research, Laguna Hills, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Oncology Specialists, SC, Park Ridge, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - McKay Urology, Charlotte, North Carolina
  - AKSM Clinical Research Group, Columbus, Ohio
  - Providence Medical Center, Portland, Oregon
  - Oregon Health and Sciences University, Portland, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - Urology Health Specialists - Bryn Mawr, Bryn Mawr, Pennsylvania
  - Albert Einstein Medical Building, Philadelphia, Pennsylvania
  - Bryn Mawr Urology Group, Rosemont, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - Urology of Virginia, PC, Virginia Beach, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beer TM, Schellhammer PF, Corman JM, Glode LM, Hall SJ, Whitmore JB, Frohlich MW, Penson DF. Quality of life after sipuleucel-T therapy: results from a randomized, double-blind study in patients with androgen-dependent prostate cancer. Urology. 2013 Aug;82(2):410-5. doi: 10.1016/j.urology.2013.04.049. PMID 23896100
- See also: USTOO International — http://www.ustoo.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Sipuleucel-T: Provenge
  Provenge: Biologic: autologous cellular product consisting of antigen presenting cells (APCs) activated with PA2024, a recombinant fusion protein composed of PAP, linked to GM-CSF
- Control: Control
  Control: Autologous cellular product consisting of antigen presenting cells (APCs) prepared in the absence of PA2024 antigen
Period: Treatment Phase 1
Arm/Group | Sipuleucel-T | Control
Started | 117 | 59
Received ≥1 Leukapherisis (Safety Set) | 116 | 59
Received ≥1 Study Product (Exposure Set) | 113 | 59
Received Booster Infusion | 50 | 30
Completed (Completed 3 scheduled infusion treatments and had confirmed Biochemical Failure (BF).) | 84 | 44
Not Completed | 33 | 15
Not completed — Disease Progression | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Patient Refused to Continue | 17 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1
Not completed — Intercurrent Illness | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 4 | 2
Not completed — Closure of Study | 3 | 2
Not completed — Completed Protocol Visits | 3 | 6
Period: Surveillance Phase
Arm/Group | Sipuleucel-T | Control
Started | 84 | 44
Completed (Reached Distant Failure (DF) following Treatment Phase.) | 41 | 13
Not Completed | 43 | 31
Not completed — Protocol Violation | 0 | 1
Not completed — Patient refused to continue | 22 | 14
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 0 | 1
Not completed — Intercurrent Illness | 2 | 0
Not completed — Other | 5 | 5
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Closure of study | 5 | 6
Not completed — Completed Protocol Visits | 3 | 2
Period: Long-term Follow-up
Arm/Group | Sipuleucel-T | Control
Started | 41 | 13
Completed (Subject survival status was assessed by phone Q6 months until death of subject. Death=Completion.) | 20 | 7
Not Completed | 21 | 6
Not completed — Patient refused to continue | 2 | 0
Not completed — Other | 5 | 0
Not completed — Closure of Study | 8 | 4
Not completed — Completed Protocol Visits | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sipuleucel-T | Control | Total
Number analyzed (Participants) | 117 | 59 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.40) | 65.2 (6.75) | 64.7 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 117 | 59 | 176
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 107 | 55 | 162
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 117 | 59 | 176
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead
  Participants
    ECOG 0=Fully Active; No restrictions. | 109 | 57 | 166
    ECOG 1= Restricted Strenuous Activity | 6 | 1 | 7
    ECOG Missing | 2 | 1 | 3
Weight [Mean (Standard Deviation); unit: Kg] | 90.45 (15.52) | 89.70 (13.85) | 90.21 (14.95)
Gleason Score [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleason Score ≤ 6 | 20 | 13 | 33
    Gleason Score =7 | 69 | 34 | 103
    Gleason Score ≥ 8 | 28 | 12 | 40
Time from diagnosis to randomization [Mean (Standard Deviation); unit: years] | 5.84 (2.76) | 6.34 (2.76) | 6.01 (2.76)

OUTCOME MEASURES:

1. Primary Outcome: Time to Biochemical Failure Cumulative Incidence Percentile
Description: Time to Biochemical Failure (TTBF) was the pre-specified primary endpoint of this trial. The biochemical failure threshold was based on evidence that prostate specific antigen (PSA) had become ≥ 3 ng/mL
Time Frame: Every 3 months post-infusion
Population: Number of subjects that met biochemical failure criteria.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sipuleucel-T | Control
Number analyzed (Participants) | 85 | 45
Months
  25th Cumulative Incidence Percentile | 7.6 [6.2 to 9.2] | 6.8 [6.1 to 9.5]
  50th Cumulative Incidence Percentile | 14.9 [9.8 to 16.1] | 12.4 [9.1 to 18.0]
  75th Cumulative Incidence Percentile | 22.9 [18.3 to 28.8] | 24.6 [17.9 to 54.0]
Statistical Analysis 1: Comparison: Sipuleucel-T vs Control; Test type: Other; p = 0.65, Log Rank; Log Rank Test (two sided) stratified by Gleason Score and Radiation Therapy; Hazard Ratio (HR) = 0.997, 95% CI 2-sided [0.693 to 1.433]

2. Primary Outcome: Number of Subjects That Met Biochemical Failure Status
Description: time to biochemical Failure (TTBF) was the pre-scpecified primary endpoint of this trial. The biochemical failure threshold was based on evidence that prostate specific antigen (PSA) had become ≥ 3 ng/mL.
Time Frame: Every 3 months post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T | Control
Number analyzed (Participants) | 117 | 59
Participants | 85 | 45

ADVERSE EVENTS:
Time Frame: AEs, regardless of relationship to product, were collected from the time of randomization through 6 months following booster administration. If the subject didn't receive a booster infusion, all AEs were collected until the time of confirmation that a booster infusion will not occur. After that time, only product related events, or any cerebrovascular event, were collected throughout the remainder of the subject's study participation (surveillance and long term follow-up study phases).
Arm/Group | Sipuleucel-T | Control
All-Cause Mortality (participants affected / at risk) | 20/116 | 9/59
Serious Adverse Events (participants affected / at risk) | 31/116 | 19/59
Other Adverse Events (participants affected / at risk) | 114/116 | 57/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=116) | Control (N=59)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (2)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 (2) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (2)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (General disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 2 (2) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ANAPLASTIC THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHRONIC MYELOMONOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 5 (6) | 3 (3)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 (1) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (2) | 1 (1)
BLADDER OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=116) | Control (N=59)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5) | 5 (6)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 3 (5) | 3 (7)
DIARRHOEA (Gastrointestinal disorders) | 14 (19) | 13 (15)
CONSTIPATION (Gastrointestinal disorders) | 16 (18) | 5 (6)
NAUSEA (Gastrointestinal disorders) | 15 (17) | 5 (6)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 8 (9) | 8 (10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 (7) | 1 (2)
FATIGUE (General disorders) | 64 (99) | 23 (36)
CHILLS (General disorders) | 51 (114) | 7 (8)
PYREXIA (General disorders) | 44 (69) | 2 (3)
INFLUENZA LIKE ILLNESS (General disorders) | 16 (23) | 3 (4)
PAIN (General disorders) | 15 (19) | 1 (1)
ASTHENIA (General disorders) | 12 (14) | 3 (7)
OEDEMA PERIPHERAL (General disorders) | 7 (8) | 7 (11)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 (25) | 7 (11)
NASOPHARYNGITIS (Infections and infestations) | 13 (15) | 7 (10)
URINARY TRACT INFECTION (Infections and infestations) | 9 (15) | 3 (5)
SINUSITIS (Infections and infestations) | 4 (7) | 4 (5)
BRONCHITIS (Infections and infestations) | 4 (5) | 3 (3)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 3 (3)
CONTUSION (Injury, poisoning and procedural complications) | 6 (7) | 7 (10)
CITRATE TOXICITY (Injury, poisoning and procedural complications) | 8 (8) | 3 (6)
WEIGHT DECREASED (Investigations) | 5 (5) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 4 (4)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 5 (5) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 29 (30) | 8 (9)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 35 (52) | 9 (9)
MYALGIA (Musculoskeletal and connective tissue disorders) | 26 (36) | 5 (8)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 9 (9) | 12 (19)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 15 (18) | 5 (5)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (6)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (5)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (8)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (6)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (9) | 3 (4)
PARAESTHESIA ORAL (Nervous system disorders) | 26 (51) | 19 (40)
HEADACHE (Nervous system disorders) | 33 (46) | 11 (17)
PARAESTHESIA (Nervous system disorders) | 21 (30) | 11 (13)
DIZZINESS (Nervous system disorders) | 14 (16) | 15 (18)
HYPOAESTHESIA (Nervous system disorders) | 5 (5) | 3 (4)
TREMOR (Nervous system disorders) | 6 (8) | 2 (4)
DEPRESSION (Psychiatric disorders) | 11 (12) | 5 (6)
INSOMNIA (Psychiatric disorders) | 13 (16) | 3 (4)
ANXIETY (Psychiatric disorders) | 9 (10) | 2 (2)
SLEEP DISORDER (Psychiatric disorders) | 4 (4) | 3 (5)
HAEMATURIA (Renal and urinary disorders) | 6 (8) | 6 (6)
DYSURIA (Renal and urinary disorders) | 5 (6) | 5 (5)
RENAL CYST (Renal and urinary disorders) | 3 (3) | 4 (4)
URINARY INCONTINENCE (Renal and urinary disorders) | 4 (4) | 6 (6)
LIBIDO DECREASED (Reproductive system and breast disorders) | 16 (16) | 14 (15)
GYNAECOMASTIA (Reproductive system and breast disorders) | 3 (3) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 5 (5)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (6)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 9 (11) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 12 (12) | 2 (2)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 8 (10) | 5 (7)
HOT FLUSH (Vascular disorders) | 78 (106) | 42 (66)
HYPERTENSION (Vascular disorders) | 17 (19) | 8 (8)
HYPOTENSION (Vascular disorders) | 7 (7) | 1 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 5 (5)
MALAISE (General disorders) | 6 (7) | 2 (2)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 4 (5) | 3 (3)
WEIGHT INCREASED (Investigations) | 7 (7) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 3 (3)
BREAST TENDERNESS (Reproductive system and breast disorders) | 1 (1) | 4 (4)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2 (2) | 3 (3)
NOCTURIA (Renal and urinary disorders) | 4 (4) | 3 (3)
AMNESIA (Nervous system disorders) | 2 (2) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 6 (7) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.